CLINICAL TRIAL: NCT05627765
Title: An Integrated Smoking Cessation and Alcohol Intervention Among Hong Kong Chinese Young People: A Feasibility Randomized Controlled Trial
Brief Title: An Integrated Smoking Cessation and Alcohol Intervention for Young People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr Eva Ho, associate professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19200161
Record Dates: First submitted 2022-04-13; First posted 2022-11-28 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Smoking Cessation; Alcohol Drinking
Keywords: Smoking cessation; Alcohol; Integrated intervention; Young adults; Feasibility; Randomized controlled trial
MeSH Terms: conditions — Smoking Cessation; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard treatment (ST) arm (Experimental): Participants will receive a brief smoking cessation intervention based on the "5A" and "5R" models proposed by the World Health Organization. The "STAR" method as quitting skills will also be provided. The "5A" model includes five steps to identify participants who are ready to quit smoking. For those who are ready to quit, a research assistant will assist them to quit using the "STAR" method: Set a quit date within 1 week, Tell the surrounding people that they have planned to quit and solicited their support, Anticipate challenges to quit attempt, and Remove all tobacco products. Otherwise, the "5R" model will be applied to those not yet ready to quit. After "5R" is applied, the research assistant will repeat the assessment of their willingness to quit. The booster interventions will be delivered by the research assistant through follow-ups arranged with the participants via phone.
  Interventions: Behavioral: Standard treatment (ST) arm
- Integrated Intervention (II) arm (Experimental): In addition to the brief smoking cessation intervention based on the "5A" and "5R" models, participants in this arm received brief advice on alcohol use based on the "FRAMES" model. The booster interventions will be delivered by the research assistant through follow-ups arranged with the participants via phone.
  Interventions: Behavioral: Integrated Intervention (II) arm
- Control arm (No Intervention): Participants will be provided with two leaflets designed by Department of health: one for smoking cessation and another for alcohol abstinence.

INTERVENTIONS:
Behavioral: Standard treatment (ST) arm — participants who are ready to quit smoking: a brief smoking cessation intervention based on the "5A" models and "STAR" method as quitting skills.
  participants who are not yet ready to quit smoking: a brief smoking cessation intervention based on the "5R" models.
  Arms: Standard treatment (ST) arm
Behavioral: Integrated Intervention (II) arm — brief advice on alcohol use based on the "FRAMES" model and the brief smoking cessation intervention based on the "5A" and "5R" models.
  Arms: Integrated Intervention (II) arm

SUMMARY:
The specific objectives of this study are to investigate the (1) feasibility, (2) preliminary effectiveness and (3) effect sizes of the integrated smoking cessation and alcohol intervention when compared to standalone smoking cessation (ST) and control among young adults in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 25 years
* smoked at least one traditional cigarette in the past 30 days
* consumed at least one alcohol unit (one "alcohol unit" contains 10g of pure alcohol) in the past 30 days
* speak Cantonese.

Exclusion Criteria:

* have a compromised mental status and/or communication problems
* participating in other smoking cessation and/or alcohol interventions

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
screening rate | From screening to the end of treatment after 6 months
  the number of smokers screened divided by the number of smokers available for screening
eligibility rate | From screening to the end of treatment after 6 months
  the number of eligible smokers divided by the number of screened people
consent rate | From screening to the end of treatment after 6 months
  the number of eligible smokers who agree to participate divided by the number of eligible smokers
randomization rate | From screening to the end of treatment after 6 months
  the number of participants who are randomized divided by the number of eligible smokers who consent to participate
attendance rate | From screening to the end of treatment after 6 months
  the number of participants who complete the intervention divided by the number of participants who are randomized into the treatment arms (ST and II)
adherence to intervention | From screening to the end of treatment after 6 months
  the number of participants in the two treatment arms who practice the skills learned during the intervention divided by the number of participants in the two treatment arms
retention rate | From screening to the end of treatment after 6 months
  the number of participants who remain in the study divided by the number of participants randomized
completion rate | From screening to the end of treatment after 6 months
  the number of participants who complete the questionnaire divided by the number of questionnaires distributed
missing data | From screening to the end of treatment after 6 months
  the percentage of missing data
adverse events | From screening to the end of treatment after 6 months
  unfavorable or unintended events during the study period that were not present at baseline or appear to have worsened since baseline

SECONDARY OUTCOMES:
Smoking quit rate | From screening to the end of treatment after 6 months
  the effect size of II on self-reported and biochemically validated quit rates for smoking at 6 months relative to ST and Control.
alcohol quit rate | From screening to the end of treatment after 6 months
  the effect size of II on self-reported quit rate for alcohol at 6 months relative to ST and Control

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yan HO, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No